CLINICAL TRIAL: NCT06854471
Title: Effects of Beverage Volume, Glycerol Concentration, and Sodium Concentration on Fluid Balance in Healthy Euhydrated Men and Women at Rest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: PEP-2420
Record Dates: First submitted 2025-02-19; First posted 2025-03-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Fluid Balance
Keywords: hydration; electrolytes; glycerol; beverage
MeSH Terms: interventions — Alkalies; Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Placebo beverage (Placebo Comparator): Base beverage, no electrolytes, no glycerol
  Interventions: Other: Placebo beverage, kiwi-strawberry flavor
- Electrolyte solution without glycerol beverage 1 (Experimental): Higher electrolytes lower volume
  Interventions: Other: Electrolyte solution without glycerol beverage 1
- Electrolyte solution without glycerol beverage 2 (Experimental): Lower electrolytes mid-volume
  Interventions: Other: Electrolyte solution without glycerol beverage 2
- Electrolyte solution without glycerol beverage 3 (Experimental): Higher electrolytes higher volume
  Interventions: Other: Electrolyte solution without glycerol beverage 3
- Electrolyte solution with glycerol beverage 1 (Experimental): Lower electrolytes, lower glycerol, lower volume
  Interventions: Other: Electrolyte solution with glycerol beverage 1
- Electrolyte solution with glycerol beverage 2 (Experimental): Higher electrolytes, higher glycerol, lower volume
  Interventions: Other: Electrolyte solution with glycerol beverage 2
- Electrolyte solution with glycerol beverage 3 (Experimental): Higher electrolytes, higher glycerol, higher volume
  Interventions: Other: Electrolyte solution with glycerol beverage 3
- Base with glycerol beverage 1 (Experimental): No electrolytes, higher glycerol, lower volume
  Interventions: Other: Base with glycerol, no electrolytes beverage 1
- Base with glycerol beverage 2 (Experimental): No electrolytes, lower glycerol, mid-volume
  Interventions: Other: Base with glycerol, no electrolytes beverage 2
- Base with glycerol beverage 3 (Experimental): No electrolytes, higher glycerol, higher volume
  Interventions: Other: Base with glycerol, no electrolytes beverage 3

INTERVENTIONS:
Other: Placebo beverage, kiwi-strawberry flavor — 9.3.oz 3 times for a total of 28 oz over a 35 min period followed by 25 min rest until Time 0 post-dose
  Arms: Placebo beverage
Other: Electrolyte solution without glycerol beverage 1 — 4 oz 3 times for a total of 12 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution without glycerol beverage 1
Other: Electrolyte solution without glycerol beverage 2 — 6.7 oz 3 times for a total of 20 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution without glycerol beverage 2
Other: Electrolyte solution without glycerol beverage 3 — 9.3.oz 3 times for a total of 28 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution without glycerol beverage 3
Other: Electrolyte solution with glycerol beverage 1 — 4 oz 3 times for a total of 12 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution with glycerol beverage 1
Other: Electrolyte solution with glycerol beverage 2 — 4 oz 3 times for a total of 12 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution with glycerol beverage 2
Other: Electrolyte solution with glycerol beverage 3 — 9.3.oz 3 times for a total of 28 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Electrolyte solution with glycerol beverage 3
Other: Base with glycerol, no electrolytes beverage 1 — 4 oz 3 times for a total of 12 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Base with glycerol beverage 1
Other: Base with glycerol, no electrolytes beverage 2 — 6.7 oz 3 times for a total of 20 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Base with glycerol beverage 2
Other: Base with glycerol, no electrolytes beverage 3 — 9.3.oz 3 times for a total of 28 oz over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: Base with glycerol beverage 3

SUMMARY:
The presence of certain ingredients such as sodium and glycerol can facilitate retention of the fluid consumed via renal water reabsorption. To maintain overall whole-body fluid balance, it is important that ingested fluid is retained in the body instead of losing it through urination.

The purpose of this study is to determine the effect of sodium and glycerol concentrations at various fluid intake volumes on fluid balance in healthy, euhydrated men and women.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant
* Subject is 18-50 years of age, inclusive
* Subject is at least recreationally active (engaged in light to moderate-intensity, intermittent, or steady-state exercise at least 3 days per week for at least 30 min at a time)
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study (e.g., diuretics)
* Subject has no health conditions that would interfere with the study (e.g. cardiovascular, renal, or metabolic diseases)
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to fast overnight (~8-12 hours)
* Subject is willing to refrain from vigorous exercise for 24 hours
* Subject is willing to eat the exact same food the day prior to each visit to the laboratory
* Provision of written consent to participate

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Fluid balance | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  Calculated as change in body mass kg and %

SECONDARY OUTCOMES:
Urine mass | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  (g)
Urine specific gravity | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  (au)
Urine osmolality | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  (mosmol/kg)
Whole blood hematocrit | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (%)
Whole blood hemoglobin concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (g/dl)
Serum sodium concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mmol/L)
Serum potassium concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mmol/L)
Serum chloride concentration (mmol/L) | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mmol/L)
Serum glucose concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mg/dl)
Serum glycerol concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mmol/L)
Serum copeptin concentration | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (pmol/L)
Serum osmolality | Change from baseline (pre-beverage) to post-beverage Time 30, 90,150 and 210 minutes
  (mosmol/kg)
Blood pressure | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  (systolic/diastolic) (mmHg)
Heart rate | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  (bpm)
Subjective measures of gastrointestinal discomfort and headache (VAS) | Change from baseline (pre-beverage) to post-beverage Time 30, 60, 90,120, 150,180 and 210 minutes
  Rated on a 100 point scale from none to severe for headache, lightheaded, stomach upset, nausea, burping, stomach bloating, abdominal discomfort, stomach fullness, vomiting, diarrhea).
Menstrual categorization | Screening visit
  Current status (e.g., contraception, regular periods or not, etc.)
Adverse Events | From Screening (Visit 1) through the fifth and final beverage testing day (Visit 6)
  Documented changes in health and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Principal Investigator — PepsiCo R&D/Gatorade and Sports Science Institute
Locations (3):
- United States (3):
  - IMG Academy/GSSI Bradenton Gatorade Sports Science Institute, Bradenton, Florida
  - GCP Research, St. Petersburg, Florida
  - Gatorade Sports Science Institute, Valhalla, New York

IPD SHARING:
Plan to Share IPD: No